CLINICAL TRIAL: NCT06148389
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-ascending Dose, Phase Ia Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Pharmacodynamics, and Immunogenicity of STSA-1301 Subcutaneous Injection in Healthy Subjects
Brief Title: The Safety and Tolerability of STSA-1301 Subcutaneous Injection in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSA-1301-01
Record Dates: First submitted 2023-10-31; First posted 2023-11-28 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2023-11

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- lowest dose group (Experimental): 4 subjects will be randomized to receive lowest dose of STSA-1301 subcutaneous injection or dose-matched placebo (First cohort)
  Interventions: Drug: STSA-1301 subcutaneous injection; Drug: Placebo
- low dose group (Experimental): 8 subjects will be randomized to receive low dose of STSA-1301 subcutaneous injection or dose-matched placebo (Second cohort)
  Interventions: Drug: STSA-1301 subcutaneous injection; Drug: Placebo
- middle dose group (Experimental): 8 subjects will be randomized to receive middle dose of STSA-1301 subcutaneous injection or dose-matched placebo (Third cohort)
  Interventions: Drug: STSA-1301 subcutaneous injection; Drug: Placebo
- high dose group (Experimental): 8 subjects will be randomized to receive high dose of STSA-1301 subcutaneous injection or dose-matched placebo (Fourth cohort)
  Interventions: Drug: STSA-1301 subcutaneous injection; Drug: Placebo
- highest dose group (Experimental): 8 subjects will be randomized to receive highest dose of STSA-1301 subcutaneous injection or dose-matched placebo (Fifth cohort)
  Interventions: Drug: STSA-1301 subcutaneous injection; Drug: Placebo

INTERVENTIONS:
Drug: STSA-1301 subcutaneous injection — Subjects will receive the administration dose on Day 0 following protocol requirements.
Drug: Placebo — Subjects will receive the administration dose on Day 0 following protocol requirements.

SUMMARY:
A randomized, double-blind, placebo-controlled, single-ascending dose, phase Ia study to evaluate the safety, tolerability, pharmacokinetic, pharmacodynamics, and immunogenicity of STSA-1301 Subcutaneous Injection in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, male and female, aged between 18 and 65 years, inclusive;
2. Body mass index: 18.0～28.0 kg/m2, inclusive; weight ≥50 kg for males and ≥45kg for females at enrollment;
3. Subjects (including their partners) agree to take highly effective contraceptive measures during the study, and they have no birth plan or sperm donation plan within 3 months after the end of the study;
4. Medical histories, physical examinations, laboratory examinations and study-related examinations and tests of the subjects show normal results or mild abnormalities with no clinical significance before enrollment, and the Investigator judges that they are eligible;
5. Subjects are aware of the risks of the study, and voluntarily participate in the clinical study and sign an informed consent form (ICF).

Exclusion Criteria:

1. Pregnant or lactating women;
2. History of cardiovascular, respiratory, kidney, liver, metabolism, endocrine, gastrointestinal, blood, nerve, skin and mental illness, cancer or other major disease that in the judgment of the Investigator might put the subject as risk on this study.
3. After splenectomy or any major surgery within 6 months prior to screening;
4. Subjects have an active infection or have a serious infection (leading to hospitalization or requiring parenteral antibiotic therapy) within 6 weeks prior to the first dose; subjects with clinically active or chronic uncontrolled bacterial, viral or fungal infections at screening;
5. Total IgG was less than the lower limit of normal at screening. Subjects with absolute neutrophil count <1.5X109/L and/or absolute lymphocyte count <1.0X109/L;
6. Subjects have a history of malignancy;
7. Subjects who are allergic to this product or any of its ingredients, history of eczema, asthma or other allergic diseases;
8. Subjects are TIGRA (T cell interferon gamma release assay) positive at screening. If TIGRA is not available, a PPD skin test may be used instead and chest imaging performed at screening showing evidence of latent/active tuberculosis (TB);
9. Positive screening test results for human immunodeficiency virus (HIV) antibodies, syphilis specific antibody, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (Anti-HCV);
10. Presence of electrocardiogram (ECG) abnormalities during the screening period, as defined by an Investigator;
11. Subjects have any conditions affecting blood collection;
12. Subjects whose daily consumption of coffee, tea and/or cola is more than 750 mL in the last 3 months before enrollment;
13. Subject who have nicotine consumption more than 5 cigarettes or the equivalent amount of tobacco per day within 3 months prior to screening;
14. Subjects whose daily consumption of alcohol at the time of screening or at any time within the prior 6 months is more than 2 standard drinks, where 1 standard drink = 360 mL or 12 oz (1 can) of regular-strength (5%) beer; 150 mL or 5 oz wine; 45 mL or 1.5 oz liquor/spirits (40%); abnormal alcohol test results at screening or baseline;
15. History of drug abuse within 1 year prior to screening; subjects with a positive urine drug abuse screen at screening or baseline;
16. Blood loss or donation>400mL within 3 months prior to screening or history of transfusion or use of any blood products within 3 months prior to enrollment;
17. Participation as a subject in any drug or vaccine or medical device clinical trial within 3 months prior to screening;
18. Vaccination or planned vaccination within 4 weeks prior to screening to 3 months after end of dosing;
19. Subjects who have taken drugs that may affect immune function within 6 months before screening, have received any monoclonal antibody or biological agent for treatment within the previous 3 months, and have previous treatment with any prescribed medications, over-the-counter (OTC) medications, herbal medicines or other supplements within 14 days prior to screening;
20. Subjects with any factors that would, in the Investigator's judgment, preclude them from participating in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Number of treatment-related adverse events as assessed by CTCAE 5.0. | 50 days
  To evaluate the safety and tolerability of STSA-1301 subcutaneous injection in healthy adult subjects.
Safety as measured by subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests. | 50 days
  Subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests (Complete Blood Count (absolute counts and %), Fasting blood glucose concentration, Serum concentrations in Electrolytes, Protein, Albumin, Total Bilirubin, Blood urea nitrogen, Creatinine, Aspartate Aminotransferase, Alanine Aminotransferase, estimated Glomerular Filtration Rate (eGFR), Activated partial thromboplastin time (aPTT), Prothrombin Time test (PT) with International Normalized Ratio (INR) and Urinalysis safety tests (pH, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, and leukocyte esterase)).
Safety as measured by subject incidence of treatment-emergent clinically significant changes in vital signs. | 50 days
  Subject incidence of treatment-emergent clinically significant changes in vital signs (Systolic and Diastolic Blood Pressure in millimeters of mercury (mmHg), Pulse Rate in beats per minute (bpm), Respiratory Rate in beats per minute (bpm) and Body temperature in Celsius).
Safety as measured by subject incidence of treatment-emergent clinically significant changes in physical examination. | 50 days
  Subject incidence of treatment-emergent clinically significant changes in physical examination (Skin mucosa, lymph nodes, head and neck, chest, abdomen, musculoskeletal, nervous system).
Safety as measured by subject incidence of treatment-emergent clinically significant changes in Electrocardiogram (ECG). | 50 days
  Subject incidence of treatment-emergent clinically significant changes in 12-lead ECGs (Heart Rate in beats per minute (bpm), PR interval in milliseconds (msec), QRS duration in milliseconds (msec), QTc in milliseconds (msec), QT interval in milliseconds (msec)).
Maximum plasma concentration (Cmax) | Pre-dose; after dose 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days and 28 days
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1301
Area under the plasma concentration-time curve from time 0 to the collection time point t of the last measurable concentration (AUC0-t) | Pre-dose; after dose 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days and 28 days
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1301
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-∞) | Pre-dose; after dose 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days and 28 days
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1301
Time of maximum concentration (Tmax) | Pre-dose; after dose 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days and 28 days
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1301
Elimination half-life (t1/2) | Pre-dose; after dose 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days and 28 days
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1301
Elimination rate constant of plasma drug concentration in terminal phase (λz) | Pre-dose; after dose 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days and 28 days
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1301
Last measurable concentration (Clast) | Pre-dose; after dose 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days and 28 days
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1301
Mean residence time (MRT) | Pre-dose; after dose 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days and 28 days
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1301
Clearance (CL) | Pre-dose; after dose 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days and 28 days
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1301
Apparent volume of distribution (Vz) | Pre-dose; after dose 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days and 28 days
  To evaluate the pharmacokinetics (PK) characteristics of STSA-1301

SECONDARY OUTCOMES:
Change from baseline in concentration of IgG. | Pre-dose; after dose 8 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days, 28 days and 49 days
  To evaluate the pharmacodynamics (PD) characteristics and immunogenicity of STSA-1301 subcutaneous injection in healthy adult subjects.
Change from baseline in concentration of anti-drug antibody | Pre-dose; after dose 14 days, 28 days, 49 days
  To evaluate the pharmacodynamics (PD) characteristics and immunogenicity of STSA-1301 subcutaneous injection in healthy adult subjects.

OTHER OUTCOMES:
Change from baseline in concentration of IgM, IgA, IgE and IgD. | Pre-dose; after dose 8 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days, 28 days and 49 days
  To evaluate the effect of STSA-1301 subcutaneous injection on Immunoglobulin, IgG subclass and cytokine.
Change from baseline in concentration of IgG1, IgG2, IgG3 and IgG4. | Pre-dose; after dose 8 hours, 24 hours, 48 hours, 72 hours, 120 hours, 168 hours, 240 hours, 14 days, 21 days, 28 days and 49 days
  To evaluate the effect of STSA-1301 subcutaneous injection on Immunoglobulin, IgG subclass and cytokine.
Change from baseline in concentration of IL-6, TNF-α. | Pre-dose; after dose 8 hours, 24 hours, 72 hours, 240 hours
  To evaluate the effect of STSA-1301 subcutaneous injection on Immunoglobulin, IgG subclass and cytokine.

CONTACTS AND LOCATIONS:
Overall Officials: Ronghua Jin, Doctor, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital,Capital Medical University, Beijing, Chaoyang District, China